CLINICAL TRIAL: NCT01991977
Title: Evaluating the Impact of 18F-DOPA-PET on Radiotherapy Planning for Newly Diagnosed Gliomas
Brief Title: 18F-DOPA-PET in Finding Tumors in Patients With Newly Diagnosed Gliomas Undergoing Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MC1374; NCI-2013-02242 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1374 (Other: Mayo Clinic); 13-005106 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-04

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — fluorodopa F 18; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (PET, pMRI, DTI, IMRT, temozolomide) (Experimental): Patients undergo 18F DOPA-PET, pMRI and DTI within 14 days before radiation therapy, 3-6 weeks after radiation therapy, and during follow-up. Patients also undergo IMRT over 30 fractions and receive temozolomide.
  Interventions: Procedure: Diffusion Weighted Imaging; Drug: Fluorine F 18 Fluorodopa; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Perfusion Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Drug: Temozolomide

INTERVENTIONS:
Procedure: Diffusion Weighted Imaging — Undergo DTI
  Other Names: Diffusion Weighted MRI; Diffusion-Weighted Magnetic Resonance Imaging; Diffusion-Weighted MR Imaging; Diffusion-Weighted MRI; DWI; DWI MRI; DWI-MRI; MR Diffusion-Weighted Imaging
Drug: Fluorine F 18 Fluorodopa — Undergo 18F-DOPA-PET
  Other Names: 18F-FDOPA
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Procedure: Perfusion Magnetic Resonance Imaging — Undergo pMRI
  Other Names: magnetic resonance perfusion imaging
Procedure: Positron Emission Tomography — Undergo 18F-DOPA-PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Temozolomide — Receive temozolomide
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This phase II trial studies how well fluorine F 18 fluorodopa (18F-DOPA)-positron emission tomography (PET) works in finding tumors in patients with newly diagnosed gliomas undergoing radiation therapy. Comparing results of diagnostic procedures done before and during radiation therapy may help doctors predict a patient's response to treatment and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare confirmed-progression free survival at 6 months for grade IV MGMT unmethylated glioma patients after radiation therapy targeting volumes designed with both 18F-DOPA PET and conventional magnetic resonance (MR) image information with historical controls from Mayo Clinic Rochester patients, including those treated on North Central Cancer Treatment Group (NCCTG) clinical trials.

SECONDARY OBJECTIVES:

I. Compare progression free survival at 12 months for grade III patients after radiation therapy targeting volumes designed with both 18F-DOPA PET and conventional MR image information with historical controls from Mayo Clinic Rochester patients, including those on NCCTG clinical trials.

II. Compare patient overall survival after radiation therapy targeting volumes designed with both 18F-DOPA PET and conventional MR image information with historical controls from Mayo Clinic Rochester patients, including those on NCCTG clinical trials.

III. Evaluate quality of life after radiotherapy treatment targeting dose escalated volumes defined to include high 18F-DOPA PET uptake.

IV. Determine acute and late effect toxicity after radiotherapy treatment targeting dose escalated volumes defined to include high 18F-DOPA PET uptake.

V. Compare confirmed-progression free survival at 12 months for grade IV MGMT methylated patients after radiation therapy targeting volumes designed with both 18F-DOPA PET and conventional MR image information with historical controls from Mayo Clinic Rochester patients, including those on NCCTG clinical trials.

VI. Compare confirmed-progression free survival in grade IV MGMT un-methylated patients with similar historical controls from Mayo Clinic Rochester patients, including those on NCCTG clinical trials.

VII. Compare confirmed-progression free survival in grade IV MGMT methylated patients with similar historical controls from Mayo Clinic Rochester patients, including those on NCCTG clinical trials.

TERTIARY OBJECTIVES:

I. Compare radiation therapy (RT) treatment volumes defined by MR only with RT treatment volumes defined with both PET and MR information for grade IV glioma patients.

II. Compare timing of accurate identification of progression defined by 18F-DOPA PET, perfusion magnetic resonance imaging (pMRI) and conventional MRI for grade IV glioma patients.

III. Compare patterns of failure after radiation therapy targeting volumes defined with target volumes designed to with both 18F-DOPA PET and conventional MR image information with patterns of failure for historical controls from Mayo Clinic Rochester patients, including those on NCCTG clinical trials.

IV. Compare RT treatment volumes defined by MR only with RT treatment volumes defined with both PET and MR information for grade III glioma patients.

V. Evaluate intra- and inter-observer variability with vs. without the addition of 18F-DOPA PET uptake for radiotherapy target volume delineation.

VI. Compare timing of accurate identification of progression defined by 18F-DOPA PET, pMRI and conventional MRI for grade III glioma patients.

VII. Compare predictive capabilities of 18F-DOPA PET, pMRI and diffusion tensor imaging (DTI) for localization of recurrences for patients treated with 18F-DOPA PET-guided RT dose escalation.

OUTLINE:

Patients undergo 18F DOPA-PET, pMRI, and DTI within 14 days before radiation therapy, 3-6 weeks after radiation therapy, and during follow-up. Patients also undergo intensity-modulated radiation therapy (IMRT) over 30 fractions and receive temozolomide.

After completion of study treatment, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed grade IV malignant glioma; Note: grade III patients are no longer being enrolled
* Computed tomography (CT) simulation, immobilization, MRI and PET imaging, treatment planning, and all follow-up MRI and PET scans to be performed at Mayo Clinic Rochester; Note: the actual radiation therapy treatments and follow-up other than imaging can be performed at Mayo Clinic Rochester, Northfield, LaCrosse, Mankato, Eau Claire, or Albert Lea
* Provide written informed consent
* Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* Patients diagnosed with anaplastic oligodendroglioma
* Unable to undergo MRI scans with contrast (e.g. cardiac pacemaker, defibrillator, kidney failure)
* Unable to undergo an 18F-DOPA PET scan (e.g. Parkinson's disease, taking anti-dopaminergic, or dopamine agonist medication or less than 6 half-lives from discontinuance of dopamine agonists); NOTE: other potentially interfering drugs consist of: amoxapine, amphetamine, benztropine, bupropion, buspirone, cocaine, mazindol, methamphetamine, methylphenidate, norephedrine, phentermine, phenylpropanolamine, selegiline, paroxetine, citalopram, and sertraline; if a patient is on any of these drugs, list which ones on the on-study form
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra H. Brinkmann, Ph.,D., Principal Investigator — Mayo Clinic in Rochester; Nadia N. Laack, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Laack NN, Pafundi D, Anderson SK, Kaufmann T, Lowe V, Hunt C, Vogen D, Yan E, Sarkaria J, Brown P, Kizilbash S, Uhm J, Ruff M, Zakhary M, Zhang Y, Seaberg M, Wan Chan Tseung HS, Kabat B, Kemp B, Brinkmann D. Initial Results of a Phase 2 Trial of 18F-DOPA PET-Guided Dose-Escalated Radiation Therapy for Glioblastoma. Int J Radiat Oncol Biol Phys. 2021 Aug 1;110(5):1383-1395. doi: 10.1016/j.ijrobp.2021.03.032. Epub 2021 Mar 23. PMID 33771703
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (PET, pMRI, DTI, IMRT, Temozolomide)
Started (Enrolled) | 91
Received PET Tracer (Received the experimental FDOPA PET tracer; evaluable for AEs) | 84
Received IMRT Treatment (Received IMRT treatment based on the FDOPA imaging results) | 79
Evaluable for the Primary Outcome (Grade IV MGMT un-methylated glioma patients after radiation therapy) | 39
Completed (Received standard of care CT simulation and received treatment) | 79
Not Completed | 12
Not completed — Withdrew prior to receiving treatment | 7
Not completed — Withdrew after start of treatment | 5

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (PET, pMRI, DTI, IMRT, Temozolomide)
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 79
  More than one race | 0
  Unknown or Not Reported | 0
Histologic grade of primary tumor [Count of Participants; unit: Participants] — Anaplastic astrocytoma (grade-III glioma) is a mid-grade tumor & diffusely infiltrating neoplasm demonstrating focal or dispersed anaplasia cells & an increased growth index compared with grade I & II astrocytoma. Pathological diagnosis is based on appearance of cells (nuclear atypia) & growth rate (mitotic activity).
  Glioblastoma (Grade-IV glioma) is the highest grade glioma tumor & is the most malignant form of astrocytoma. The histologic features include: presence of necrosis (dead cells), increase of abnormal growth of blood vessels around the tumor, tumors are always rapidly growing.
  Participants
    Grade 3 | 4
    Grade 4 | 75
MGMT [Count of Participants; unit: Participants] — MGMT : O6-methylguanine-DNA methyltransferase methylation status
  PET : Positron-emission tomography
  pMRI : parallel magnetic resonance imaging
  DTI : Diffusion Tensor Imaging
  IMRT : Intensity-modulated radiation therapy
  Participants
    Methylated | 25
    Un-Methylated | 39
    NA | 15

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Grade IV MGMT Un-methylated Patients That Experience Confirmed-progression-free Survival at 6 Months (CPFS6)
Description: The proportion of Grade IV MGMT un-methylated patients that experience confirmed-progression-free survival at 6 months (CPFS6). Progression is defined by any of the following:
  * ≥25% increase in the sum of products of perpendicular diameters of enhancing lesions compared to the smallest tumor measurement obtained either at baseline or best response, on stable or increasing doses of corticosteroids
  * Significant increase in T2/FLAIR non-enhancing lesion on stable or increasing doses of corticosteroids compared to baseline scan or best response following initiation of therapy, not due to co-morbid events
  * Any new lesion
  * Clear clinical deterioration not attributable to other causes apart from the tumor or changes in corticosteroid dose.
  * Failure to return for evaluation due to death or deteriorating condition
  * Clear progression of non-measurable disease
Time Frame: Time from registration to the confirmed disease progression, assessed at 6 months
Population: All Grade IV MGMT un-methylated patients meeting eligibility criteria who have signed a consent form and who have begun treatment with 18F-DOPA PET image-guided dose escalation RT will be evaluable for the endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Diagnostic (PET, pMRI, DTI, IMRT, Temozolomide)
Number analyzed (Participants) | 39
proportion of participants | 0.795 [0.631 to 0.901]

2. Secondary Outcome: Overall Survival
Description: The median survival time and 95%CI will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Population: All eligible patients were included in analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Diagnostic (PET, pMRI, DTI, IMRT, Temozolomide)
Number analyzed (Participants) | 63
months
  Unmethylated patients: number analyzed (Participants) | 39
  Unmethylated patients | 16.0 [13.8 to 21.1]
  Methylated patients: number analyzed (Participants) | 24
  Methylated patients | 35.5 [25.5 to 74.4]

3. Secondary Outcome: Progression Free Survival
Description: The median progression-free survival time and 95%CI will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Population: All patients eligible for analysis were included
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Diagnostic (PET, pMRI, DTI, IMRT, Temozolomide)
Number analyzed (Participants) | 63
months
  Unmethylated patients: number analyzed (Participants) | 39
  Unmethylated patients | 8.7 [7.6 to 11.0]
  Methylated patients: number analyzed (Participants) | 24
  Methylated patients | 10.7 [8.9 to 16.0]

4. Secondary Outcome: Quality of Life Evaluated With the M. D. Anderson Symptom Inventory - Brain Tumor (MDASI-BT) Questionnaire
Description: The MDASI-BT consists of 28 questions. Twenty-two questions are related to severity of symptoms over the last 24 hours and are answered on a scale of 0-10 where 0=not present and10=as bad as you can imagine. The remaining 6 questions are related to how symptoms have interfered with daily life over the past 24 hours and are answered on a scale of 0-10 where 0=did not interfere and 10=interfered completely. Higher scores indicate greater severity of symptoms and greater interference with daily life. Analysis will include median change percent from baseline.
Time Frame: Up to 5 years
Population: Patients that completed an assessment at baseline and at the first MRI assessment were included in analysis
Measure: Median (Full Range); unit: percent change
Arm/Group | Diagnostic (PET, pMRI, DTI, IMRT, Temozolomide)
Number analyzed (Participants) | 61
percent change | -0.167 [-6.3 to 8.17]

5. Secondary Outcome: Number of Patients Experiencing Grade 3+ Treatment-related Toxicities
Description: Adverse events graded using Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (PET, pMRI, DTI, IMRT, Temozolomide)
Number analyzed (Participants) | 75
Participants | 17

6. Secondary Outcome: Number of Patients Experiencing Grade 4+ Late Treatment-related Toxicities
Description: Late treatment-related toxicities will be assessed using the Radiation Therapy Oncology Group (RTOG) European Organization for Research and the Treatment of Cancer (EORTC) toxicity criteria.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (PET, pMRI, DTI, IMRT, Temozolomide)
Number analyzed (Participants) | 63
Participants | 0

7. Other Pre Specified Outcome: Inter-observer Variability With or Without the Addition of 18F-DOPA Positron Emission Tomography Uptake for Radiotherapy Target Volume Delineation
Description: The concordance correlation coefficient will be used to measure agreement between volumes generated with each method, as well as to evaluate inter-observer variability, where variability associated with magnetic resonance imaging will serve as the standard for comparison.
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Intra-observer Variability With or Without the Addition of 18F-DOPA Positron Emission Tomography Uptake for Radiotherapy Target Volume Delineation
Description: as for outcome 7
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Magnetic Resonance Imaging-only Defined Volumes and the Volumes Defined With the Combination of Magnetic Resonance and Positron Emission Tomography Planning
Description: Paired t-test statistical analysis will be performed to determine if any differences exist and the level of statistical significance between treatment volumes defined by magnetic resonance imaging only and treatment volumes defined with both positron emission tomography and magnetic resonance imaging information. The analysis of volumes from 72 grade IV patients will have 90% power to detect differences in volumes with an effect size of 0.39 using a paired t-test with a 0.05 two-sided significance level. Alternate metrics for comparison will also be assessed, including spatial overlap, distanc
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Patterns of Failure After Radiation Therapy Targeting Volumes by 18F-DOPA Positron Emission Tomography and Conventional Magnetic Resonance Imaging
Description: Chi-square tests of proportions will be used to test for differences in the proportions of patients with central, in-field, marginal, or distant failures between the patients on this study and historical controls.
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Predictive Capabilities of 18F-DOPA Positron Emission Tomography, Perfusion Magnetic Resonance Imaging, and Diffusion Tensor Imaging for Localization of Recurrences
Description: Compared by identifying the recurrence volume with each modality and correlating with identification of aggressive disease in the pre-radiation therapy planning images.
Time Frame: Up to 5 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Radiation Therapy Treatment Volumes Defined by Magnetic Resonance Imaging Only and Defined With Both Positron Emission Tomography and Magnetic Resonance Imaging Information for Grade III Glioma Patients
Description: Paired t-test statistical analysis will be performed to determine if any differences exist and the level of statistical significance between treatment volumes defined by magnetic resonance imaging only and treatment volumes defined with both positron emission tomography and magnetic resonance imaging information.
Time Frame: Up to 5 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Radiation Therapy Treatment Volumes Defined by Magnetic Resonance Imaging Only or Defined With Both Positron Emission Tomography and Magnetic Resonance Imaging Information for Grade IV Glioma Patients
Description: Paired t-test statistical analysis will be performed to determine if any differences exist and the level of statistical significance between treatment volumes defined by magnetic resonance imaging only and treatment volumes defined with both positron emission tomography and magnetic resonance imaging information. The analysis of volumes from 72 grade IV patients will have 90% power to detect differences in volumes with an effect size of 0.39 using a paired t-test with a 0.05 two-sided significance level. Alternate metrics for comparison will also be assessed, including spatial overlap, distan
Time Frame: Up to 5 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Timing of Accurate Identification of Progression Defined by 18F- DOPA Positron Emission Tomography, Perfusion Magnetic Resonance Imaging and Conventional Magnetic Resonance Imaging for Grade IV Glioma Patients
Description: The progression identification timing will be compared by calculating the percentage of time each modality was earlier than conventional magnetic resonance imaging. With a sample size of 72, if the observed percentage earlier than conventional magnetic resonance imaging is 30% for either modality, a two-sided 95% confidence interval for a single proportion using the large sample normal approximation will be +/- 10.6%. Progression identification timing will also be compared using Kaplan-Meier methods and paired t-tests to determine if differences exist between the modalities.
Time Frame: Up to 5 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Timing of Accurate Identification of Progression Defined by 18F- DOPA Positron Emission Tomography, Perfusion Magnetic Resonance Imaging and Conventional Magnetic Resonance Imaging for Grade III Glioma Patients
Description: Progression identification timing will be compared using Kaplan-Meier methods and paired t-tests to determine if differences exist between the modalities. An exploratory analysis of diffusion tensor imaging for detecting invasive non-enhancing tumor recurrence will also be performed.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Diagnostic (PET, pMRI, DTI, IMRT, Temozolomide)
All-Cause Mortality (participants affected / at risk) | 56/84
Serious Adverse Events (participants affected / at risk) | 3/84
Other Adverse Events (participants affected / at risk) | 82/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (PET, pMRI, DTI, IMRT, Temozolomide) (N=84)
Fatigue (General disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (PET, pMRI, DTI, IMRT, Temozolomide) (N=84)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (2)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (2)
Endocrine disorders - Other, specify (Endocrine disorders) | 2 (2)
Blurred vision (Eye disorders) | 3 (4)
Eye disorders - Other, specify (Eye disorders) | 2 (2)
Optic nerve disorder (Eye disorders) | 1 (2)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (5)
Fatigue (General disorders) | 81 (329)
Fever (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 2 (4)
Upper respiratory infection (Infections and infestations) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 4 (4)
Platelet count decreased (Investigations) | 3 (3)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 6 (7)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 3 (5)
Central nervous system necrosis (Nervous system disorders) | 28 (81)
Cognitive disturbance (Nervous system disorders) | 9 (14)
Concentration impairment (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 4 (6)
Dysphasia (Nervous system disorders) | 5 (5)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 12 (14)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 5 (7)
Muscle weakness left-sided (Nervous system disorders) | 6 (9)
Muscle weakness right-sided (Nervous system disorders) | 4 (5)
Nervous system disorders - Oth spec (Nervous system disorders) | 10 (19)
Neuralgia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 9 (11)
Somnolence (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (21)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT01991977/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT01991977/ICF_001.pdf